CLINICAL TRIAL: NCT05285371
Title: Intravenous Hydration After Surgery Using Boluses of Balanced Salt Solution
Brief Title: Boluses of Ringer's in Surgical Kids (BRiSK Study)
Acronym: BRiSK
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-019180
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dehydration in Children; Fluid Therapy
Keywords: Hydration; Fluids; Lactated Ringer's; Hyponatremia; Dehydration; Post Operative; Pediatrics; Children; Intravenous Fluid Therapy
MeSH Terms: conditions — Hyponatremia; Dehydration | interventions — Urinalysis

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized into one of two groups - Continuous (CONT) or Bolus (BOL).
  CONT group will receive traditional continuous D50.45% NaCl + 20 mEq/L KCl solution at 2/3 maintenance rate.
  BOL group will receive intravenous boluses of Lactated Ringer's at 2/3-maintenance rate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CONT Group (Placebo Comparator): CONT group will receive standard traditional intravenous fluid of D50.45% NaCl + 20 mEq/L KCl at 2/3 maintenance rate.
  Interventions: Diagnostic Test: Urinalysis (UA); Diagnostic Test: Complete Metabolic Panel (CMP); Diagnostic Test: Glucose Stick Test (d-Stick); Other: Medical Chart Review
- BOL Group (Experimental): BOL group will receive intravenous boluses of Lactated Ringer's three times daily at 2/3 maintenance rate.
  Interventions: Diagnostic Test: Urinalysis (UA); Diagnostic Test: Complete Metabolic Panel (CMP); Diagnostic Test: Glucose Stick Test (d-Stick); Other: Medical Chart Review

INTERVENTIONS:
Diagnostic Test: Urinalysis (UA) — Urinalysis will be performed twice daily starting on Postoperative Day 0.
Diagnostic Test: Complete Metabolic Panel (CMP) — A CMP will be performed on Postoperative Day 2 and Postoperative Day 4.
Diagnostic Test: Glucose Stick Test (d-Stick) — A d-Stick will be performed twice daily except on Postoperative Day 2 and Postoperative Day 4 as the CMP includes serum glucose levels.
Other: Medical Chart Review — A medical chart review will be performed for all subjects enrolled.

SUMMARY:
Traditional protocols for intravenous fluid administration in children who have undergone a major abdominal or thoracic operation are based on a landmark paper published in 1957 by Holliday and Segar. The basic tenets include: (1) Continuous intravenous fluid administration; (2) Total fluid volume based on the "4:2:1" rule; (3) Use of hypotonic electrolyte solutions, most commonly 0.45% sodium chloride (NaCl) + 20 milliequivalents per liter (mEq/L) potassium chloride (KCl); and (4) Inclusion of 5% dextrose to increase the osmolarity of the infusate and to help prevent ketosis and acidemia.

DETAILED DESCRIPTION:
Recent studies have questioned the validity of each of these tenets. Maintenance rate as defined by Holliday & Segar is postulated to be in excess of pediatric patients' post-surgical fluid needs. The investigators propose a novel protocol for the administration of IV fluids to children after major abdominal or thoracic surgery that includes: (1) Intermittent boluses; (2) Total volume administered in 24 hours closer to 2/3 of the traditional maintenance fluid requirements; and (3) Use of a balanced salt solution (Lactated Ringer).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 12 months to 21 years.
2. Weight >= 8 kg.
3. Patients with an uncomplicated abdominal or thoracic surgical procedure in which the expected postoperative length of stay is anticipated to be at least 2-5 days.
4. Patients admitted to a regular bed following surgery.
5. Patients who will be inpatient for approximately 4-8 days postoperatively.
6. Parental/guardian permission (informed consent).

Exclusion Criteria:

1. Patients with a history of diabetes, seizures, hyperglycemia, and hypoglycemia.
2. Patients prescribed insulin.
3. Patients receiving parenteral nutrition.
4. Patients with excessive GI losses (small bowel obstruction, severe diarrhea, large-volume ascites or drainage).
5. Complicated surgery that requires an ICU or ICU transfer immediately after surgery.
6. Patients with any form of hypersensitivity to the study fluids.
7. Laboratory abnormalities that indicate clinically significant hematologic, hepatobiliary, or renal disease:

   * Serum Sodium <130 or >145 mmol/L
   * Serum Potassium <3.0 or >5.0 mEq/L
   * Serum Chloride <90 or >110 mEq/L
   * Serum Creatinine ≥ 1.6 mg/dL
   * Serum Glucose <60 or >180 mg/dL
   * Alanine Aminotransferase >200 U/L
   * Total Bilirubin >12.0 mg/dL
8. Pregnant or lactating females.
9. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Fluid Adherence to Study Protocol | 4 Days
  Feasibility will be determined if 85% of enrolled study participants receive at least 75% of the expected study fluid in accordance to study protocol.
Feasibility of Measuring and Collecting Urine Output | 4 Days
  Feasibility will be determined if at least 90% of enrolled study participants have accurate urine collection and urine measurements during the study treatment phase.

SECONDARY OUTCOMES:
Feasibility of Study Laboratory Tests - CMP, d-Stick, Urinalysis | 4 Days
  Feasibility will be determined if at least 70% of enrolled study participants have at least 75% of study laboratory tests collected and recorded during the study treatment phase.
Feasibility of Randomization | Baseline
  Feasibility will be determined if at least 85% of eligible study participants are subsequently enrolled, consented, and randomized during their pre-operative phase of care.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mattei, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] McNab S. Intravenous maintenance fluid therapy in children. J Paediatr Child Health. 2016 Feb;52(2):137-40. doi: 10.1111/jpc.13076. PMID 27062616
- [Background] Rooholamini SN, Clifton H, Haaland W, McGrath C, Vora SB, Crowell CS, Romero H, Foti J. Outcomes of a Clinical Pathway to Standardize Use of Maintenance Intravenous Fluids. Hosp Pediatr. 2017 Dec;7(12):703-709. doi: 10.1542/hpeds.2017-0099. PMID 29162640
- [Background] Neville KA, Sandeman DJ, Rubinstein A, Henry GM, McGlynn M, Walker JL. Prevention of hyponatremia during maintenance intravenous fluid administration: a prospective randomized study of fluid type versus fluid rate. J Pediatr. 2010 Feb;156(2):313-9.e1-2. doi: 10.1016/j.jpeds.2009.07.059. Epub 2009 Oct 9. PMID 19818450
- [Background] Bagri NK, Saurabh VK, Basu S, Kumar A. Isotonic versus Hypotonic Intravenous Maintenance Fluids in Children: A Randomized Controlled Trial. Indian J Pediatr. 2019 Nov;86(11):1011-1016. doi: 10.1007/s12098-019-03011-5. Epub 2019 Jul 6. PMID 31280410
- [Background] Morgan JA. Question 2: Should 0.9% saline be used for maintenance fluids in hospitalised children? Arch Dis Child. 2015 Jul;100(7):715-7. doi: 10.1136/archdischild-2015-308821. Epub 2015 May 20. No abstract available. PMID 25994003
- [Background] Moritz ML. Syndrome of Inappropriate Antidiuresis. Pediatr Clin North Am. 2019 Feb;66(1):209-226. doi: 10.1016/j.pcl.2018.09.005. PMID 30454744
- [Background] Feld LG, Neuspiel DR, Foster BA, Leu MG, Garber MD, Austin K, Basu RK, Conway EE Jr, Fehr JJ, Hawkins C, Kaplan RL, Rowe EV, Waseem M, Moritz ML; SUBCOMMITTEE ON FLUID AND ELECTROLYTE THERAPY. Clinical Practice Guideline: Maintenance Intravenous Fluids in Children. Pediatrics. 2018 Dec;142(6):e20183083. doi: 10.1542/peds.2018-3083. PMID 30478247
- [Background] Friedman JN, Beck CE, DeGroot J, Geary DF, Sklansky DJ, Freedman SB. Comparison of isotonic and hypotonic intravenous maintenance fluids: a randomized clinical trial. JAMA Pediatr. 2015 May;169(5):445-51. doi: 10.1001/jamapediatrics.2014.3809. PMID 25751673
- [Background] Moritz ML, Ayus JC. Hospital-acquired hyponatremia--why are hypotonic parenteral fluids still being used? Nat Clin Pract Nephrol. 2007 Jul;3(7):374-82. doi: 10.1038/ncpneph0526. PMID 17592470
- [Background] Oh GJ, Sutherland SM. Perioperative fluid management and postoperative hyponatremia in children. Pediatr Nephrol. 2016 Jan;31(1):53-60. doi: 10.1007/s00467-015-3081-y. Epub 2015 Mar 18. PMID 25784018
- [Background] Abdessalam S. Hypotonic versus isotonic maintenance fluid administration in the pediatric surgical patient. Semin Pediatr Surg. 2019 Feb;28(1):43-46. doi: 10.1053/j.sempedsurg.2019.01.007. Epub 2019 Jan 23. PMID 30824133
- [Background] McNab S, Ware RS, Neville KA, Choong K, Coulthard MG, Duke T, Davidson A, Dorofaeff T. Isotonic versus hypotonic solutions for maintenance intravenous fluid administration in children. Cochrane Database Syst Rev. 2014 Dec 18;2014(12):CD009457. doi: 10.1002/14651858.CD009457.pub2. PMID 25519949
- [Background] Easley D, Tillman E. Hospital-acquired hyponatremia in pediatric patients: a review of the literature. J Pediatr Pharmacol Ther. 2013 Apr;18(2):105-11. doi: 10.5863/1551-6776-18.2.105. PMID 23798904
- [Background] Moritz ML, Ayus JC. Prevention of hospital-acquired hyponatremia: a case for using isotonic saline. Pediatrics. 2003 Feb;111(2):227-30. doi: 10.1542/peds.111.2.227. PMID 12563043
- [Background] Malbrain MLNG, Langer T, Annane D, Gattinoni L, Elbers P, Hahn RG, De Laet I, Minini A, Wong A, Ince C, Muckart D, Mythen M, Caironi P, Van Regenmortel N. Intravenous fluid therapy in the perioperative and critical care setting: Executive summary of the International Fluid Academy (IFA). Ann Intensive Care. 2020 May 24;10(1):64. doi: 10.1186/s13613-020-00679-3. PMID 32449147
- [Background] Bampoe S, Odor PM, Dushianthan A, Bennett-Guerrero E, Cro S, Gan TJ, Grocott MP, James MF, Mythen MG, O'Malley CM, Roche AM, Rowan K, Burdett E. Perioperative administration of buffered versus non-buffered crystalloid intravenous fluid to improve outcomes following adult surgical procedures. Cochrane Database Syst Rev. 2017 Sep 21;9(9):CD004089. doi: 10.1002/14651858.CD004089.pub3. PMID 28933805
- [Background] Chin KJ, Macachor J, Ong KC, Ong BC. A comparison of 5% dextrose in 0.9% normal saline versus non-dextrose-containing crystalloids as the initial intravenous replacement fluid in elective surgery. Anaesth Intensive Care. 2006 Oct;34(5):613-7. doi: 10.1177/0310057X0603400511. PMID 17061636
- [Background] Self WH, Semler MW, Wanderer JP, Wang L, Byrne DW, Collins SP, Slovis CM, Lindsell CJ, Ehrenfeld JM, Siew ED, Shaw AD, Bernard GR, Rice TW; SALT-ED Investigators. Balanced Crystalloids versus Saline in Noncritically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):819-828. doi: 10.1056/NEJMoa1711586. Epub 2018 Feb 27. PMID 29485926
- [Background] Maheshwari K, Turan A, Makarova N, Ma C, Esa WAS, Ruetzler K, Barsoum S, Kuhel AG, Ritchey MR, Higuera-Rueda C, Kopyeva T, Stocchi L, Essber H, Cohen B, Suleiman I, Bajracharya GR, Chelnick D, Mascha EJ, Kurz A, Sessler DI. Saline versus Lactated Ringer's Solution: The Saline or Lactated Ringer's (SOLAR) Trial. Anesthesiology. 2020 Apr;132(4):614-624. doi: 10.1097/ALN.0000000000003130. PMID 31977517
- [Background] Farrell PR, Farrell LM, Hornung L, Abu-El-Haija M. Use of Lactated Ringers Solution Compared With Normal Saline Is Associated With Shorter Length of Stay in Pediatric Acute Pancreatitis. Pancreas. 2020 Mar;49(3):375-380. doi: 10.1097/MPA.0000000000001498. PMID 32132512